CLINICAL TRIAL: NCT06429488
Title: Obsessive-compulsive Disorder, Depression and Anxiety Among Patients With Crohn's Disease
Status: Completed | Type: Observational
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Mohammad Sami El Muhtaseb, Associate Professor, University of Jordan
Other Study IDs: 233/2022
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- chron's disease patients: patients diagnosed with CD at the department of Gastroenterology were collected from hospital records, and all patients were contacted and accepted to be part of this study
  Interventions: Other: no intervention, questionnaires were used
- Healthy controls: Healthy Controls with no medical illness or mental illness before were invited to fill in the same questionnaire, the controls were relatives of patients attending the hospital for clinics not related to the gastrointestinal tract or psychiatry
  Interventions: Other: no intervention, questionnaires were used

INTERVENTIONS:
Other: no intervention, questionnaires were used — The following psychological assessment tools were used:
  Obsessive-Compulsive Inventory-Revised (OCI-R): An 18-item self-report questionnaire measuring symptoms across six subscales: washing, checking, neutralizing, obsessing, ordering, and hoarding. A score of 21 or higher indicates likely OCD.
  Depression Anxiety Stress Scales-21 (DASS-21): A set of three self-report scales assessing stress, depression, and anxiety over 21 items. This shortened version is widely used for research and clinical purposes and is easy to administer.
  Patient Health Questionnaire-9 (PHQ-9): A nine-item scale for assessing depressive symptoms. Scores are categorized as: 1-4 (no/minimal), 5-9 (mild), 10-14 (moderate), 15-19 (moderately severe), and 20-27 (severe depression).
  Generalized Anxiety Disorder-7 (GAD-7): A seven-item tool measuring anxiety symptoms and the severity of generalized anxiety disorder (GAD).

SUMMARY:
Introduction: Crohn's disease (CD) and obsessive-compulsive disorder (OCD) are two distinct medical conditions that affect millions of people worldwide. While numerous studies have explored anxiety and depression in CD, there is a notable lack of research about the link between OCD and CD. The aim of the study is to look for a relation between these seemingly unrelated conditions.

Methods: Patients with a diagnosis of Crohn's disease were given four different questionnaires in order to assess for the presence of obsessive-compulsive disorder, depression, and anxiety symptoms using the OCI-R score, DASS-21, PHQ-9, and GAD-7. The same questionnaires were used to assess healthy controls for similar symptoms.

DETAILED DESCRIPTION:
This is an observational case-control study conducted at Jordan University Hospital. Using hospital medical records, patients with Crohn's disease who had been treated and followed up at the gastro-enterology and colorectal clinics were contacted to obtain consent to participate in the research and to explain its goals and the nature of the questionnaires used. Patients who agreed to participate were sent an online questionnaire to fill in. Healthy Controls with no medical illness or mental illness were invited to fill in the same questionnaire. The controls were relatives of patients attending the hospital for clinics not related to the gastrointestinal tract or psychiatry. Patients and controls with documented psychiatric illnesses were excluded.

The following psychological assessment tools were used:

The Obsessive-Compulsive Inventory-Revised (OCI-R) for obsessive-compulsive symptoms. It is composed of an 18-item self-report validated questionnaire that measures symptoms across 6 subscales including washing, checking, neutralizing, obsessing, ordering, and hoarding. The possible range of scores is 0-72.

The Depression Anxiety Stress Scales-21 (DASS-21) for overall emotional well-being. It is a set of three self-report scales to understand the degree of stress and distress, depressive and anxiety symptoms. The shortened version was used, which consists of 21 items and has been widely used for research and clinical purposes and is easy to administer.

The Patient Health Questionnaire-9 (PHQ-9), a nine-item depression scale of the patient health questionnaire, to assess depressive symptoms. The individual responses are interpreted as a score, with depression divided from no depression to severe depression.

The Generalized Anxiety Disorder-7 (GAD-7), a seven-item tool used to measure or assess anxiety symptoms and the severity of generalized anxiety disorder (GAD).

Data analysis:

The data was collected using Microsoft Forms and downloaded into Excel for coding and deidentification before being imported into the Statistical Package for Social Science (IBM SPSS Statistics for Windows, version 25, IBM Corp., Armonk, N.Y., USA) for analysis. The chi-square test was used to compare different categorical variables. The Mann-Whitney U test was used to compare non-categorical variables. The Kruskal-Wallis test was applied to test for significant differences between the scales.

Ethical consideration:

This study adhered to the principles of the Declaration of Helsinki 1975 and was approved by the Institutional Review Board at Jordan University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Crohn's disease who have been treated and followed up at the gastro-enterology and colorectal clinics of Jordan University Hospital.
* Patients who have provided informed consent to participate in the research after being informed about the study's goals and the nature of the questionnaires used.
* Healthy controls with no prior history of medical or mental illness.
* Controls who are relatives of patients attending non-gastroenterology and non-psychiatry clinics at Jordan University Hospital.
* Participants (both patients and healthy controls) who agree to fill in the online questionnaire.

Exclusion Criteria:

- Patients and controls with documented psychiatric illnesses.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This is an observational case-control study was conducted at Jordan University Hospital, Using hospital medical records, patients with Crohn's disease who been treated and followed up at the gastro-enterology and colorectal clinics were contacted to obtain their consent to participate in the research and to explain its goals and the nature of the questionnaires used. Patients who agreed to participate were sent an online questionnaire to fill in. Healthy Controls with no medical illness or mental illness before were invited to fill in the same questionnaire, the controls where relatives of patients attending the hospital for clinics not related to the gastrointestinal tract or psychiatry. Patients and controls with documented psychiatric illnesses were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 293 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
This study aims to determine the prevalence of obsessive-compulsive disorder in patients with CD and compare it with people without CD (controls) | 6 months
  The Depression Anxiety Stress Scales-21 (DASS-21)

SECONDARY OUTCOMES:
This study aims to determine the Patient Health Questionnaire-9 (PHQ-9) in patients with CD and compare it with people without CD (controls) | 6 months
  The Patient Health Questionnaire-9 (PHQ-9)
This study aims to determine the Generalized Anxiety Disorder-7 (GAD-7) in patients with CD and compare it with people without CD (controls) | 6 months
  The Generalized Anxiety Disorder-7 (GAD-7)

CONTACTS AND LOCATIONS:
Locations (1):
- the Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No